CLINICAL TRIAL: NCT05154734
Title: Efficacy and Safety of Belimumab in Neuromyelitis Optica Spectrum Disorders (BEAT NMO)
Brief Title: Efficacy and Safety of Belimumab in Neuromyelitis Optica Spectrum Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Department of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2021-YX-187-01
Record Dates: First submitted 2021-12-07; First posted 2021-12-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — belimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belimumab (Experimental): Belimumab will be intravenously administered with a dose of 10mg/kg on Days 0,14 and28, then every 28 days until week 48, with a final evaluation at week 52.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab will be intravenously administered with a dose of 10mg/kg on Days 0,14 and28, then every 28 days until week 48, with a final evaluation at week 52.

SUMMARY:
Neuromyelitis Optica Spectrum Disorders (NMOSD) is associated with a pathological humoral immune response against the aquaporin-4(AQP-4) water channel. Belimumab (Benlysta ®) is a human immunoglobulin G1λ monoclonal antibody that inhibits B-cell survival and differentiation by neutralizing soluble B lymphocyte stimulator. Belimumab may benefit some patients with NMOSD due to the important role of B cells in the pathogenesis of NMOSD. Clinical trials may be needed to observe its efficacy and safety.

DETAILED DESCRIPTION:
The investigators primarily aim to observe the number of attacks from initiation of belimumab treatment.

The secondary outcomes are to determine: The safety profile of belimumab in participants with NMO and whether belimumab improves Expanded Disability Status Scale (EDSS), et al.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old
2. Diagnosis of NMO or NMO spectrum disorder according to the 2015 International Panel for Neuromyelitis Optica Diagnosis criteria
3. Clinical evidence of either at least one attack requiring rescue therapy (intravenous corticosteroids, intravenous immunoglobulin, plasma exchange, or a combination of these therapies) in the year before screening or at least two attacks requiring rescue therapy in the 2 years before screening.
4. EDSS <= 6.0
5. Patients were seropositive for AQP4-IgG
6. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection (Herpes simplex virus, varicella-zoster virus, cytomegalovirus, Epstein-Barr virus, human immunodeficiency virus, Hepatitis viruses, Syphilis, etc)
2. Participation in another interventional trial within the last 3 months
3. Tumor disease currently or within last 5 years
4. Pregnant, breastfeeding, or child-bearing potential during the course of the study
5. Clinically relevant heart, liver, kidney or bone marrow function disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
The number of attacks | From baseline to one year after
  An acute attack was defined as a new neurological worsening lasting for at least 24 hours and occurring more than 30 days after the previous attack.

SECONDARY OUTCOMES:
Worsening in EDSS | Worsening from baseline in EDSS to 52 weeks
  The Expanded Disability Status Scale (EDSS) is a rating system that is frequently used for classifying and standardizing the severity and progression. EDSS ranges from 0 to 10.
Number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Optic nerve,brain and spinal cord Magnetic Resonance Imaging (MRI) | From baseline to 52 weeks
  The total number of new and/or enlarging T2 lesions for all participants was calculated as the sum of the individual number of lesions at Weeks 12, 24, and 52
Counts of peripheral blood B cell subsets | From baseline to 52 weeks
  Compare peripheral blood plasma cells before and one year after initial intervention
Determination of serum AQP4 antibodies | From baseline to 52 weeks
  Compare serum AQP4-ab titers before and one year after initial intervention
Incidence of treatment-emergent adverse events [safety and tolerability] | From baseline to 52 weeks
  Adverse events related to belimumab are recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China